CLINICAL TRIAL: NCT05868603
Title: Effect of Different Remineralization Gels on the White Spot Lesions
Brief Title: Effect of Different Remineralization Gels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haner Direskeneli, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: müdf.24.04.23
Record Dates: First submitted 2023-04-24; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remineralization gel with CPP- ACP (GC Tooth MousseTM, Tokyo, Japan) (Experimental): CPP-ACP containing remineralization gel (Tooth Mousse GC, Tokyo, Japan) will be put into the Essix appliance with a reservoir and applied for 5-7 minutes twice a day for one month.
  Before and after the applying remineralization gel, the laser fluorescence values will measure with a DIAGNOdent pen (KaVo Dental corporation, East Main street Lake Zurich, lL).
  Interventions: Other: Remineralization gel
- Remineralization gel with calcium glycerophosphate (R.O.C.S.® Medical Mineral Gel, Russia) (Experimental): Remineralization gel containing calcium glycerophosphate (R.O.C.S.® Medical Minerals Gel, Russia) will be put into the Essix appliance with a reservoir for 5-7 minutes twice a day for one month. Before and after the applying remineralization gel, the laser fluorescence values will measure with a DIAGNOdent pen( KaVo Dental corporation, East Main street Lake Zurich, lL).
  Interventions: Other: Remineralization gel
- Control Group (No Intervention): No intervention.

INTERVENTIONS:
Other: Remineralization gel — Remineralization gel
  Arms: Remineralization gel with CPP- ACP (GC Tooth MousseTM, Tokyo, Japan); Remineralization gel with calcium glycerophosphate (R.O.C.S.® Medical Mineral Gel, Russia)

SUMMARY:
The aim of the study is to treat white spot lesions that occur after orthodontic treatment.

Different gels will be used for remineralization. The study will consist of 45 people between the ages of 15-18. 45 people will be divided into 3 groups.

DETAILED DESCRIPTION:
Oral hygiene training will be given to each group and a toothpaste containing 1450 ppm fluoride will be given to brush their teeth twice a day.

Essix appliance with reservoir will be made by taking impressions from 30 patients. Remineralization gel will be put into the Essix appliance for 5-7 minutes twice a day for one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-18 years,
* Presence of white point lesions,
* Volunteering to participate in the research.

Exclusion Criteria:

* Not having received orthodontic treatment,
* Having a developmental anomaly affecting the enamel,
* Being allergic to milk,
* Having a syndrome affecting the oral cavity.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-24 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) | 4 weeks
  Decrease in laser fluorescence values with Diagnodent Pen as an indicator of remineralization

SECONDARY OUTCOMES:
Calcium glycerophosphate | 4 weeks
  Decrease in laser fluorescence values with Diagnodent Pen as an indicator of remineralization

IPD SHARING:
Plan to Share IPD: No